CLINICAL TRIAL: NCT05416801
Title: Investigation of University Level Volleyball Players in Terms of Ankle Functions and Postural Control Variables
Status: Completed | Type: Observational
Sponsor: Istanbul Gelisim University (Other)
Collaborators: Yeditepe University (Other)
Responsible Party: Principal Investigator, Aysem Ecem Ozdemir, Research Assistant, Istanbul Gelisim University
Other Study IDs: YU001
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Volleyball; Ankle; Postural Balance
Keywords: postural control; ankle; range of motion; strenght; vibration; proprioception; volleyball

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Volleyball Group: Female Volleyball players who are currently playing in a university team and who are meeting the inclusion criteria.
- Control Group: Female university students who are meeting the inclusion criteria.

SUMMARY:
In this study, it is aimed to evaluate different ankle functions and postural control variables in university level volleyball players and students with stable ankles and to examine the results obtained. In this way, we aim to contribute to the physiotherapy and rehabilitation literature and clinical studies of physiotherapists who are interested in athlete health.

The hypothesis set in this study is:

H0: There is no difference between ankle functions and postural control variables of volleyball players and healthy controls.

H1: There is a difference between ankle functions and postural control variables of volleyball players and healthy controls.

DETAILED DESCRIPTION:
There are studies proving that athletes with poor postural control have a higher risk of injury to the ankle and knee regions than those with normal. Balanced stance and effective postural control in activities involving ball contact during the game are the basic skills of volleyball. The ankle is a joint that needs to be evaluated frequently and its functions should be improved both in order to improve postural control ability and to prevent possible injuries. It has been proven in studies that the capacity shown in different functional parameters such as joint range of motion, strength and proprioception and balance both reduces the risk of injury and positively reflects on the performance parameters of the athlete. It will be useful to evaluate and examine the ankle functions and postural controls that change as a result of the training and exercises performed by the athletes, unlike healthy individuals who are not athletes, in order to understand the abilities developed specifically for the sport.

The study will be carried out in Yeditepe University Physiotherapy and Rehabilitation Graduate Laboratory. Female individuals aged 18-25 years, with stable ankles will be included in the study as a sample. The study will consist of two groups. The first group will include volleyball players playing in university teams, and healthy university students meeting the same criteria in the control group. The sample size of the study was calculated using the GPower program as type 1 error value= 0.05, power = 0.90, effect size (f value) calculated from the reference article and total of 40 subjects for the independent sample t-test.

The Cumberland Ankle Instability Tool will be used to select suitable participants for the study. Only ankles considered stable according to the questionnaire will be included in this study. First, static balance will be evaluated with the PK Prokin 252 system during the silent stand for postural control assessment. Then, different ankle functions of the people who will participate in the study will be evaluated. The measurement of the range of motion of the ankle will be evaluated with the help of a goniometer. Different degrees of position sense of the ankle joint will be evaluated with the aid of a goniometer and the sense of vibration will be evaluated with a tuning fork. Muscle strength will be measured with the help of a manual dynamometer during the movements of the muscles around the ankle. In addition, the participants who volunteered to participate in the study before the tests will be given a Voluntary Consent Form and a Demographic Information Form. Participants will be given rest periods between each test. Evaluation time will be 45 minutes for each participant. Participants will not be followed up after the assessments.

ELIGIBILITY:
Inclusion Criteria:

* Female gender,
* Being between the ages of 18-25,
* Having a score of ≥24 on the Cumberland Ankle Instability Questionnaire,
* Volunteering for the study.

Exclusion Criteria:

* Presence of neuromuscular system disease,
* Presence of vestibular or visual problems,
* Presence of acute or chronic pain,
* An ankle injury in the last year,
* For the control group, regular participation in sports activities or physical activity for more than 150 minutes, 5 days a week.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study was carried out with female individuals aged 18-25 who have stable ankles and have not had an ankle injury in the last 1 year. The study includes volleyball players playing in university teams and healthy university students who meet the same criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Postural control | Baseline
  Postural control is evaluated according to the results of the static stability test performed on the PK Prokin 252 balance device with proven reliability. Postural control outcome is measured by the findings of the Prokin System, wich are: Average center of gravity on the X-axis (mm), Average Y-axis center of gravity (mm), Forward-backward standard deviation (mm), Medial-lateral standard deviation (mm) variables.
Ankle Joint Range of Motion | Baseline
  Range of motion assessment is made using a goniometer. Dorsiflexion and plantarflexion in the tibiotalar joint, and eversion and inversion in the subtalar joint is evaluated both actively and passivley. These evaluations will be repeated 3 times and their averages will be recorded.
Ankle Joint Proprioception | Baseline
  The assessment is made by a goniometer. First the referance degree is passively tought and then while eyes are closed, the person tries to reach the referance degree. The movements starts from 145 degrees of plantar flexion to the degrees of 105, 120, 130 and 140.
Vibration Sense | Baseline
  Vibration evaluation is made with the help of tuning fork (128 Hz). The eyes are closed throughout the application. Reference points are the big toe, fifth toe, and medial malleolus. The person is instructed to say when the feeling of vibration ends. A timer was used to count the time.
Ankle Joint Muscle Strength | Baseline
  The maximum isometric strength of the ankle is evaluated with the manual dynamometer measurement, the validity and reliability of which has been proven. JTECH Commander Powertrack Manual Dynamometer was used for measurements. Dorsiflexion, plantar flexion, eversion and inversion movements are assessed.

OTHER OUTCOMES:
Cumberland Ankle Instability Tool | Baseline
  The tool is used to to understand if the ankle is stable or unstable. The scale consists of nine questions about ankle joint functions and whether there is pain in different activities and a total of 30 points. Functional instability increases with low scores from the questionnaire. The cutoff point for the stable ankle is ≥24.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No